CLINICAL TRIAL: NCT05046535
Title: The Effect of Cigarette Smoke on Sleep Quality and Physical Activity in People With Multiple Sclerosis
Acronym: Smoke-MS
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Mayis Aldughmi, Associate Professor, University of Jordan
Other Study IDs: 2021-2020/26
Record Dates: First submitted 2021-09-05; First posted 2021-09-16 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis
Keywords: Sleep quality; Cigarette Smoking; Physical Activity; Secondhand smoke
MeSH Terms: conditions — Multiple Sclerosis; Sleep Initiation and Maintenance Disorders; Cigarette Smoking; Motor Activity | interventions — Exercise; Nicotine Chewing Gum; Smoking Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA sequencing for 20-25 subjects out of the whole sample will be performed. Sanger sequencing to all subjects will also be performed to identify related genes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smokers: Individuals with MS who are current tobacco smokers: Either cigarettes, hookah pipe, E-cigarettes or other forms of tobacco. This group will perform all the assessments including surveys about nicotine dependence and smoking behavior.
  Interventions: Behavioral: Sleep quality and physical activity; Genetic: Nicotine dependence; Diagnostic Test: Nicotine and cotinine serum levels; Behavioral: Smoking
- Non-smokers: Individuals with MS who are non-smokers of any form of tobacco. This group will perform all the assessments except for the surveys related to nicotine dependence and smoking behavior.
  Interventions: Behavioral: Sleep quality and physical activity; Diagnostic Test: Nicotine and cotinine serum levels

INTERVENTIONS:
Behavioral: Sleep quality and physical activity — Self-reported assessments will be used to measure the following: overall sleep quality, insomnia symptoms, Obstructive sleep apnea.
  Physical activity will be measured objectively using the 6MWT, 9HPT, and cardiorespiratory fitness using the VO2 submaximal test on the recumbent stepper.
Genetic: Nicotine dependence — DNA sequencing for 20-25 subjects out of the whole sample will be performed. Sanger sequencing to all subjects will also be performed to identify related genes
  Groups: Smokers
Diagnostic Test: Nicotine and cotinine serum levels — Cotinine serum level which is a major metabolite of nicotine and the preferred biomarker for measuring tobacco use will be measured together with nicotine levels using Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS).
Behavioral: Smoking — Surveys that measure nicotine dependence and smoking behavior
  Groups: Smokers

SUMMARY:
Current evidence suggests that cigarette smoke increases disease progression in people with multiple sclerosis (PwMS) and worsen their symptoms. 70% of PwMS report sleep disturbances that negatively affects their quality of life. Cigarette smoke has been found to be associated with sleep disturbances in healthy adult smokers, but this relationship is unknown in PwMS. Also, those who smoke cigarettes have less physical endurance resulting in undesirable effects on physical activity. Also, current evidence suggests that genes play a major role in smoking behavior and that certain genetic differences greatly affects nicotine dependence. To our knowledge, this was never explored before among PwMS.

This study aims to explore the association between cigarette smoke, sleep quality, and physical activity in PwMS. Another aim is to explore the genetic susceptibility of people with MS to cigarette smoke, specifically to nicotine dependence

DETAILED DESCRIPTION:
Prevalence of Cigarette Smoke in Jordan

29% of the adult population in Jordan are smokers, making it the highest rate in the middle east. According to the 2017 WHO report, smoking prevalence is increasing in the eastern Mediterranean region, in which Jordan is the leading country across the middle east with the worst ratings in cigarette smoke. Another recent study in 2019 conducted by the Jordanian government in collaboration with the WHO, showed that eight out of ten men in Jordan regularly smoke nicotine and consume around 23 cigarettes per day. Therefore, the percentage of Jordanian men who smoke increased up to 66% and 17% for Jordanian women, making these rates dangerously high.

Impact of Cigarette Smoke

Cigarette smoke accounts for six million deaths annually worldwide and is a major cause of morbidity, increasing the risk of developing cancer, cardiovascular disease, and pulmonary infections. Cigarette smoke has been found to be associated with sleep disturbances in healthy adult smokers. In addition, those who smoke cigarettes have less physical endurance and performance, decreased muscle strength and flexibility affecting their overall physical fitness and health.

Nicotine in cigarette smoke may disrupt sleep quality through several mechanisms. The release of neurotransmitters that disrupts the normal sleep-wake cycle such as dopamine and serotonin, disruption in the circadian rhythms that may develop chronic conditions such as depression, and craving nicotine during the night due to nicotine dependence may all disrupts a cigarette smoker night of sleep. Carbon monoxide and other toxins found in cigarette smoke affects the binding of oxygen to red blood cells affecting the delivery of oxygen to active muscles, heart, and lungs which might explain the low physical fitness level of smokers.

Sleep Quality in Multiple Sclerosis

Multiple Sclerosis (MS) is a neurodegenerative disease characterized by the destruction of myelin in the central nervous system. People with MS often present with a variety of symptoms including sleep disturbances that affects around 70 % of these individuals. Sleep disorders such as obstructive sleep apnea and insomnia are also commonly seen among this population. Poor sleep quality affect people with MS daily physical function, and may worsen other symptoms such as depression, pain, and fatigue. Sleep disturbances in MS may be due to primary factors that result from lesions in brain areas controlling sleep/wake cycles, or secondary factors which are due to medication side-effects or symptoms that accompany MS such as pain, fatigue, depression, and bowl and bladder problems.

Smoking and Multiple Sclerosis

Research in the area of cigarette smoke and MS suggests that smoking increases the risk of developing MS, increase the number of relapses and disease severity among people with MS, fasten their transfer into more progressive forms, reduce the effectiveness of their disease-modifying therapies, and worsen symptoms such as pain, motor deficits, and cognitive impairments. It is suggested that cigarette smoke alter the immune response and induce inflammatory changes in people with MS which might explain the host of negative effects it has on MS disease status.

Genetics and Smoking

Current evidence suggests that genes play a major role in smoking behavior and that certain genetic differences greatly affects nicotine dependence among healthy individuals. These genes can ultimately affect how an individual initiate and quit smoking. There is also evidence that showed specific genes are associated with an increased risk of developing smoking related diseases such as cardiovascular diseases. Therefore, it would be interesting to explore genetic predisposition to nicotine dependence among PwMS. Understanding the effect of genes on cigarette smoke behavior will greatly influence the decision making on effective smoking cessation treatments in the future.

Significance of Study

As current evidence from the healthy smoking population suggests those who smoke cigarettes have more sleep disturbances compared to non-smokers, people with MS who smoke cigarettes may have poorer sleep quality and higher risk of developing sleep disorders such as obstructive sleep apnea. In addition, being physical inactive negatively influence the rehabilitation process of people with MS. It affects their participation in therapy and can result in deconditioning of their muscles and joints worsening their symptoms. It can also affect other quality of life indices including their social interpersonal relationships and employment rates. Despite the evidence on the effects of cigarette smoke in people with MS, to our knowledge, no previous study has explored the relationship between smoking status, sleep quality, and physical activity in people with MS.

Considering the high prevalence of cigarette smoke in Jordan and its negative effects on the overall well-being of individuals specially people with MS, It is crucial to explore its relationship with common symptoms among a sample of Jordanian people with MS. Another area of this project that the researchers are interested to explore is the genetic susceptibility of people with MS to cigarette smoke, specifically to nicotine dependence.

Although this has been studied before in health smokers, no previous study has explored this among people with MS. Understanding the role genes play on smoking behavior among PwMS will guide future large scale studies to further explore this relationship and eventually provide guidance to smoking cessation programs.

The researchers of this project believe that findings from this study will:

1. Shed the light on a major public health problem and its association with health-related outcomes in PwMS.
2. Increase awareness on the negative effects of cigarette smoke among PwMS, health-care providers, and researchers.
3. Increase awareness on the importance of physical activity among PwMS as well as health care providers to promote physical activity among their clients.
4. Shed the light on the important effect of the genomic material on the behaviors of adults which will influence cigarette smoke treatment and prevention options
5. Provide the base for future studies to explore management options such as smoking cessation programs and physical activity for the aim to improve sleep quality in PwMS.
6. Generate recommendations among health care providers to promote sleep health among PwMS and policy makers to enforce stricter regulations on promoting, using, and selling cigarettes in Jordan and the World.

ELIGIBILITY:
Inclusion Criteria

1. Confirmed diagnosis of MS from a neurologist using the McDonald diagnostic criteria
2. Ability to ambulate independently with or without an assistive device
3. Current, previous, and nonsmokers
4. Age ≥ 18 years
5. Ability to give informed consent.

Exclusion Criteria

1. A neurological disease other than MS
2. Orthopedic problems or other conditions that may significantly interfere with testing
3. Uncorrected vision loss
4. Acute ischemic cardiovascular event or coronary artery bypass surgery less than 3 months ago
5. Uncontrolled blood pressure with medication (BP>190/110mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with MS who are current or non smokers and who are able to ambulate independently with or without an assistive device
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Nicotine and cotinine serum levels | 6 months
  Cotinine serum level which is a major metabolite of nicotine and the preferred biomarker for measuring tobacco use will be measured together with nicotine levels using Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS). Analysis of serum cotinine and nicotine levels will be performed in collaboration with Smart Labs group which is a certified external medical laboratory and the only facility in Jordan that analyze serum nicotine levels. Blood samples will be collected and stored at the CTC then transferred to Smart Labs for analyses.
Sleep quality | 6 months
  Sleep quality will be assessed subjectively using the following surveys which are validated in PwMS and are available in Arabic language: Pittsburgh Sleep Quality Index that assess global sleep quality, Epworth Sleepiness Scale that assess daytime sleepiness, Insomnia Severity Index that assess the risk of having insomnia, and STOP-Bang questionnaire that assesses the risk of having obstructive sleep apnea.
Physical activity and cardiorespiratory fitness | 6 months
  Physical activity will be assessed subjectively using the International Physical Activity Questionnaire, and objectively using the 6-Minute Walk Test which is a measure of physical performance and endurance. Maximum Volume of Oxygen consumption (VO2 Max) which is a measure of cardiorespiratory fitness will be quantified using the submaximal test on the recumbent stepper machine.

SECONDARY OUTCOMES:
Genetic predisposition to nicotine dependence and other blood tests | 6 months
  DNA sequencing for 20-25 subjects out of the whole sample will be performed. Sanger sequencing to all subjects will also be performed to identify related genes. ELISA oxidative stress microarray will also be performed to all subjects. Vitamin D levels will also be detected from the subject's blood sample. Blood samples will be collected, stored, and analyzed at the CTC.

OTHER OUTCOMES:
Depression | 6 months
  depression will be measured using the Beck Depression Inventory (BDI)
Fatigue | 6 months
  Fatigue will be measured using the Modified Fatigue Impact Scale (MFIS)
Manual dexterity | 6 months
  Upper extremity function will be measured using the Nine-hole peg test (9HPT) which is a test that measures upper extremity manual dexterity
Cognitive function | 6 months
  The Montreal Cognitive Assessment (MoCA) will be used to assess global cognitive function. The Symbol Digits Modalities Test (SDMT) will be utilized to assess information processing speed (Most affected cognitive domain in MS).

CONTACTS AND LOCATIONS:
Overall Officials: Mayis Aldughmi, PhD, Principal Investigator — University of Jordan
Locations (1):
- Cell Therapy Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hedstrom AK, Olsson T, Alfredsson L. Smoking is a major preventable risk factor for multiple sclerosis. Mult Scler. 2016 Jul;22(8):1021-6. doi: 10.1177/1352458515609794. Epub 2015 Oct 12. PMID 26459151
- [Background] Correale J, Farez MF. Smoking worsens multiple sclerosis prognosis: two different pathways are involved. J Neuroimmunol. 2015 Apr 15;281:23-34. doi: 10.1016/j.jneuroim.2015.03.006. Epub 2015 Mar 6. PMID 25867464
- [Background] Alrouji M, Manouchehrinia A, Gran B, Constantinescu CS. Effects of cigarette smoke on immunity, neuroinflammation and multiple sclerosis. J Neuroimmunol. 2019 Apr 15;329:24-34. doi: 10.1016/j.jneuroim.2018.10.004. Epub 2018 Oct 9. PMID 30361070
- [Background] Braley TJ, Chervin RD. A practical approach to the diagnosis and management of sleep disorders in patients with multiple sclerosis. Ther Adv Neurol Disord. 2015 Nov;8(6):294-310. doi: 10.1177/1756285615605698. PMID 26600873
- [Background] Purani H, Friedrichsen S, Allen AM. Sleep quality in cigarette smokers: Associations with smoking-related outcomes and exercise. Addict Behav. 2019 Mar;90:71-76. doi: 10.1016/j.addbeh.2018.10.023. Epub 2018 Oct 17. PMID 30368021
- [Background] Dugas EN, Sylvestre MP, O'Loughlin EK, Brunet J, Kakinami L, Constantin E, O'Loughlin J. Nicotine dependence and sleep quality in young adults. Addict Behav. 2017 Feb;65:154-160. doi: 10.1016/j.addbeh.2016.10.020. Epub 2016 Oct 25. PMID 27816041
- [Background] Chen LJ, Steptoe A, Chen YH, Ku PW, Lin CH. Physical activity, smoking, and the incidence of clinically diagnosed insomnia. Sleep Med. 2017 Feb;30:189-194. doi: 10.1016/j.sleep.2016.06.040. Epub 2016 Nov 25. PMID 28215247
- [Background] Veauthier C, Paul F. Sleep disorders in multiple sclerosis and their relationship to fatigue. Sleep Med. 2014 Jan;15(1):5-14. doi: 10.1016/j.sleep.2013.08.791. Epub 2013 Nov 15. PMID 24360534
- [Background] Jaehne A, Unbehaun T, Feige B, Lutz UC, Batra A, Riemann D. How smoking affects sleep: a polysomnographical analysis. Sleep Med. 2012 Dec;13(10):1286-92. doi: 10.1016/j.sleep.2012.06.026. Epub 2012 Sep 28. PMID 23026505
- [Background] Newland P, Flick L, Salter A, Dixon D, Jensen MP. The link between smoking status and co-morbid conditions in individuals with multiple sclerosis (MS). Disabil Health J. 2017 Oct;10(4):587-591. doi: 10.1016/j.dhjo.2017.03.005. Epub 2017 Mar 23. PMID 28351749
- [Background] Ozcan ME, Ince B, Bingol A, Erturk S, Altinoz MA, Karadeli HH, Kocer A, Asil T. Association between smoking and cognitive impairment in multiple sclerosis. Neuropsychiatr Dis Treat. 2014 Sep 10;10:1715-9. doi: 10.2147/NDT.S68389. eCollection 2014. PMID 25246792
- [Background] El-Salem K, Al-Shimmery E, Horany K, Al-Refai A, Al-Hayk K, Khader Y. Multiple sclerosis in Jordan: A clinical and epidemiological study. J Neurol. 2006 Sep;253(9):1210-6. doi: 10.1007/s00415-006-0203-2. Epub 2006 Apr 28. PMID 16649096
- [Background] Manouchehrinia A, Weston M, Tench CR, Britton J, Constantinescu CS. Tobacco smoking and excess mortality in multiple sclerosis: a cohort study. J Neurol Neurosurg Psychiatry. 2014 Oct;85(10):1091-5. doi: 10.1136/jnnp-2013-307187. Epub 2014 Feb 25. PMID 24569687
- [Background] Raja M, Garg A, Yadav P, Jha K, Handa S. Diagnostic Methods for Detection of Cotinine Level in Tobacco Users: A Review. J Clin Diagn Res. 2016 Mar;10(3):ZE04-6. doi: 10.7860/JCDR/2016/17360.7423. Epub 2016 Mar 1. PMID 27135020
- [Background] Davies GE, Soundy TJ. The genetics of smoking and nicotine addiction. S D Med. 2009;Spec No:43-9. PMID 19363894
- [Background] Domingue BW, Conley D, Fletcher J, Boardman JD. Cohort Effects in the Genetic Influence on Smoking. Behav Genet. 2016 Jan;46(1):31-42. doi: 10.1007/s10519-015-9731-9. Epub 2015 Jul 30. PMID 26223473